CLINICAL TRIAL: NCT05067894
Title: A Phase I, Observer-Blind, Randomized, Controlled Study of the Safety and Immunogenicity of SARS-CoV-2 Protein Subunit Recombinant Vaccine in Healthy Populations Aged 18 Years and Above in Indonesia
Brief Title: Safety and Immunogenicity of SARS-CoV-2 Protein Subunit Recombinant Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Collaborators: Fakultas Kedokteran Universitas Indonesia (Other); National Institute of Health Research and Development, Ministry of Health Republic of Indonesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CoV2-010221
Record Dates: First submitted 2021-10-01; First posted 2021-10-05 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Covid19
Keywords: covid19 vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Observer blind: Investigational Product and Active Comparator are masking. Lot number is masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Adult - Vaccine candidate (Experimental): 50 µg dose, adult group (18-59 years)
  Interventions: Biological: SARS-CoV-2 Protein Subunit Recombinant Vaccine
- Adult - Control (Active Comparator): SARS-CoV-2 inactivated vaccine, adult group (18-59 years)
  Interventions: Biological: SARS-CoV-2 Inactivated Vaccine
- Elderly - Vaccine candidate (Experimental): 50 µg dose, elderly group (> 60 years)
  Interventions: Biological: SARS-CoV-2 Protein Subunit Recombinant Vaccine
- Elderly - Control (Active Comparator): SARS-CoV-2 inactivated vaccine, elderly group (> 60 years)
  Interventions: Biological: SARS-CoV-2 Inactivated Vaccine

INTERVENTIONS:
Biological: SARS-CoV-2 Protein Subunit Recombinant Vaccine — intramuscular injection
  Arms: Adult - Vaccine candidate; Elderly - Vaccine candidate
Biological: SARS-CoV-2 Inactivated Vaccine — intramuscular injection
  Arms: Adult - Control; Elderly - Control

SUMMARY:
The study is an observer-blind, randomized, controlled prospective intervention study of Phase I. The primary objective is To evaluate the safety of the SARS-CoV-2 protein subunit recombinant vaccine within 7 days after each dose.

DETAILED DESCRIPTION:
This trial is observer blinded, comparative, randomized, phase I study. Approximately 60 subjects will be recruited (18 years and above).

The investigational product is 0.5 ml in three dose-regimen (for all subjects) with 28 days apart between doses, compare to an active control (inactivated SARS-CoV-2 vaccine)

ELIGIBILITY:
Inclusion Criteria:

1. Clinically healthy subjects within the following age groups: adults (18-59 years) and elderly (60 years and above.
2. Subjects have been informed properly regarding the study and signed the informed consent form.
3. Subjects will commit to comply with the instructions of the investigator and the schedule of the trial.

Exclusion Criteria:

1. Subjects concomitantly enrolled or scheduled to be enrolled in another trial.
2. History of vaccination with any investigational product against Covid-19 during or 6 months prior to enrollment.
3. Subjects who have history of Covid-19 in the last 3 months (based on anamnesis or other examinations).
4. Evolving mild, moderate or severe illness, especially infectious disease or fever (body temperature ≥37.5℃, measured with infrared thermometer/thermal gun).
5. The result of rapid antigen test is positive.
6. Women who are lactating, pregnant or planning to become pregnant during the study period (judged by self-report of subjects and urine pregnancy test results).
7. Abnormality hematology and biochemical test results.
8. History of asthma, history of allergy to vaccines or vaccine ingredients, and severe adverse reactions to vaccines, such as urticaria, dyspnea, and angioneurotic edema.
9. History of uncontrolled coagulopathy or blood disorders contraindicating intramuscular injection.
10. Patients with serious chronic diseases (serious cardiovascular diseases, uncontrolled hypertension and diabetes, liver and kidney diseases, malignant tumors, etc) which according to the investigator might interfere with the assessment of the trial objectives.
11. Subjects who have any history of confirmed or suspected immunosuppressive or immunodeficient state, or received in the previous 4 weeks a treatment likely to alter the immune response (intravenous immunoglobulins, blood-derived products or long-term corticosteroid therapy (> 2 weeks)).
12. Subjects who have history of uncontrolled epilepsy or other progressive neurological disorders, such as Guillain-Barre Syndrome.
13. Subjects receive any vaccination (other than Covid-19 vaccine) within 1 month before and after Investigational Product (IP) immunization.
14. Subjects plan to move from the study area before the end of study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-08-06 (Actual)

PRIMARY OUTCOMES:
Safety of the SARS-CoV-2 protein subunit recombinant vaccine within 7 days after each dose | 7 days after each dose
  percentage of subjects with solicited and unsolicited Adverse Events (AE)

SECONDARY OUTCOMES:
safety of the SARS-CoV-2 protein subunit recombinant vaccine within 28 days after each dose | 28 days after each dose
  percentage of subjects with solicited and unsolicited AE
Comparison of AE/ Serious Adverse Events (SAE) between intervention vaccine and active control | 28 days after each dose
  percentage of subjects with AE and SAE between vaccine and active control group
Deviation of laboratory evaluation | 28 days after the first dose
  Any deviation from routine laboratory evaluation that probably related to the dosing
Deviation of laboratory evaluation | 7 days after whole schedule dose
  Any deviation from routine laboratory evaluation that probably related to the dosing
Immunogenicity profile of the SARS-CoV-2 protein subunit recombinant vaccine after second dose | 28 days after each dose
  seropositive rate, seroconversion rate and GMT of IgG antibody and neutralization antibody
Comparison of immunogenicity between 2 and 3 doses | 28 days after second and third dose
  seropositive rate, seroconversion rate and GMT of IgG antibody and neutralization antibody

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Rini Sekartini, MD, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- Fakultas Kedokteran Universitas Indonesia, Jakarta, Greater Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No